CLINICAL TRIAL: NCT04278417
Title: A 96-week, Two-arm, Randomized, Single-masked, Multi-center, Phase III Study Assessing the Efficacy and Safety of Brolucizumab 6 mg Compared to Panretinal Photocoagulation Laser in Patients With Proliferative Diabetic Retinopathy
Brief Title: Study of Efficacy and Safety of Brolucizumab Versus Panretinal Photocoagulation Laser in Patients With Proliferative Diabetic Retinopathy
Acronym: CONDOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRTH258D2301
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: proliferative diabetic retinophathy, retinal neovascularization, anti-VEGF, brolucizumab, intravitreal injection, panretinal photocoagulation
MeSH Terms: conditions — Retinal Neovascularization | interventions — brolucizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): Intra-vitreal injection. 3 x q6w loading injections, followed by q12w maintenance through Week 90
  Interventions: Biological: Brolucizumab 6 mg
- Panretinal photocoagulation laser Arm (Active Comparator): Initial treatment in 1-4 sessions up to Week 12, followed with additional PRP treatment as needed
  Interventions: Procedure: Panretinal photocoagulation laser

INTERVENTIONS:
Biological: Brolucizumab 6 mg — 3 x q6w loading injections, followed by q12w maintenance through Week 90
  Other Names: RTH258
  Arms: Brolucizumab 6 mg
Procedure: Panretinal photocoagulation laser — initial treatment in 1-4 sessions up to Week 12, followed with additional PRP treatment as needed
  Other Names: PRP
  Arms: Panretinal photocoagulation laser Arm

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of brolucizumab compared to panretinal photocoagulation laser (PRP) in patients with proliferative diabetic retinopathy (PDR). This evaluation will provide information that brolucizumab is non-inferior to PRP with respect to the change in best corrected visual acuity at Week 54.

DETAILED DESCRIPTION:
Phase III, 96-week, two-arm, randomized (1:1 ratio), single-masked, multi-center, active-controlled study to evaluate the efficacy and safety of brolucizumab compared to Panretinal photocoagulation (PRP) in subjects with Proliferative diabetic retinopathy (PDR).

Subjects who consented underwent screening assessments to evaluate their eligibility based on the inclusion and exclusion criteria. Subjects who met all the inclusion and none of the exclusion criteria were randomized in a 1:1 ratio to one of the following treatments:

Brolucizumab 6 mg: 3 x q6w loading then q12w maintenance through Week 90, with the option from Week 48 onwards to extend the treatment interval by 6 weeks at a time up to 24 weeks, and revert to q12w if disease worsens. More frequent injection with q6w interval in the maintenance phase could be administered at the discretion of the Investigator if the disease worsens.

PRP: initial treatment in 1-4 sessions up to Week 12, followed with additional PRP treatment (may split into 2-4 sessions) as needed up to Week 90.

Visits occurred every 6 weeks throughout the study, regardless of treatment or not.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation
* Able to complete adequate fundus photographs and retinal images
* Diagnosis of type 1 or 2 Diabetes Mellitus (DM) and HbA1c less than or equal to 12% at screening
* DM treatment stable for at least 3 months
* PDR diagnosis with no previous PRP treatment in the study eye

Exclusion Criteria:

* Concomitant conditions or ocular disorders in the study eye at Screening or Baseline that could compromise a response to study treatment.
* Presence of diabetic macular edema in the study eye
* Active infection or inflammation in the study eye
* Uncontrolled glaucoma (IOP greater than 25 mmHg)
* Intravitreal anti-VEGF treatment within 6 months
* Treatment with intraocular corticosteroids
* End stage renal disease requiring dialysis or kidney transplant
* Uncontrolled blood pressure
* Systemic anti-VEGF therapy at any time

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (114):
- United States (40):
  - Retina Associates SW, Tucson, Arizona
  - Retina- Vitreous Assoc Medical Group, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - Salehi Retina Institute, Huntington Beach, California
  - Retina Consultants of Southern California, Redlands, California
  - Premiere Practice Management LLC, Torrance, California
  - Lundquist Inst BioMed at Harbor, Torrance, California
  - Miramar Eye Specialists, Ventura, California
  - Advanced Research LLC, Deerfield Beach, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - Pinnacle Research Institute, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Retina Institute, Jacksonville, Florida
  - Blue Oc Clin Res at Palm Bch Eye Ct, Lakeland, Florida
  - MedEye Associates, Miami, Florida
  - Florida Retina Institute, Orlando, Florida
  - Eye Center of North Florida, Panama City, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Associates, Elmhurst, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - John-Kenyon American Eye Institute PC, New Albany, Indiana
  - Retina Associates PA, Lenexa, Kansas
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - University of Mississippi Med Ctr, Jackson, Mississippi
  - Retina Associates Of Cleveland, Cleveland, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Cascade Medical Research Institute, Springfield, Oregon
  - Erie Retinal Surgery, Erie, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Southeastern Retina Associates P C, Knoxville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Texan Eye P A, Austin, Texas
  - Retina And Vitreous Of Texas, Bellaire, Texas
  - Retina Consultants TX Rsrch Ctr, Bellaire, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Valley Retina Institute PA, Harlingen, Texas
  - Retina Consultants of Houston PA, Houston, Texas
  - Medical Center Opthamology Assoc, San Antonio, Texas
  - Retina Associates Of South Texas PA, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
- Argentina (4):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Rosario, De Santa Fe
  - Novartis Investigative Site, CABA
- Australia (4):
  - Novartis Investigative Site, Albury, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Strathfield, New South Wales
- Brazil (4):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sorocaba, São Paulo
- Canada (4):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Boisbriand, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Novartis Investigative Site, Santiago, RM, Chile
- China (13):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xi'an, Shaanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- India (5):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Tirunelveli, Tamil Nadu
  - Novartis Investigative Site, Chandigarh
  - Novartis Investigative Site, New Delhi
- Japan (17):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sakura, Chiba
  - Novartis Investigative Site, Yoshida-gun, Fukui
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Kobe
  - Novartis Investigative Site, Osaka
- Mexico (3):
  - Novartis Investigative Site, Ciudad de, Mexico City
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Tijuana
- Philippines (3):
  - Novartis Investigative Site, Makati, NCR
  - Novartis Investigative Site, Makati
  - Novartis Investigative Site, Pasig
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico
- Russia (6):
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Sterlitamak
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Yekaterinburg
- South Korea (4):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Hualien City
  - Novartis Investigative Site, Kaohsiung City
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2680

RESULTS

PARTICIPANT FLOW:
Groups:
- Brolucizumab 6 mg: Brolucizumab 6 mg: 3 x q6w loading then q12w maintenance through Week 90, with the option from Week 48 onwards to extend the treatment interval by 6 weeks at a time up to 24 weeks and revert to q12w if disease worsens. More frequent injection with q6w interval in the maintenance phase could be administered at the discretion of the Investigator if the disease worsens.
- Panretinal Photocoagulation Laser Arm: Initial treatment in 1-4 sessions up to Week 12, followed by additional PRP treatment as needed.
Period: Overall Study
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Started | 347 | 342
Completed | 301 | 287
Not Completed | 46 | 55
Not completed — Withdrawal by Subject | 20 | 20
Not completed — Progressive disease | 0 | 2
Not completed — Physician Decision | 4 | 6
Not completed — Lost to Follow-up | 11 | 13
Not completed — Death | 8 | 9
Not completed — Adverse Event | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm | Total
Number analyzed (Participants) | 347 | 342 | 689
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (11.88) | 54.7 (10.83) | 53.9 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 132 | 276
  Male | 203 | 210 | 413
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 157 | 148 | 305
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 5
  Black or African American | 22 | 16 | 38
  White | 166 | 169 | 335
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) at Week 54 for the Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of >= 34 ETDRS letters (Snellen equivalent 20/200) at Screening / Baseline in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better functioning.
  Last observation carried forward (LOCF) was used for the imputation of missing values.
Time Frame: Baseline, Week 54
Population: Full Analysis Set- Last Observation Carried Forward (FAS - LOCF), for patients with a valid measurement with no protocol deviations with impact.
Measure: Least Squares Mean (Standard Error); unit: Letters Read
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 342 | 337
Letters Read | 0.2 (0.72) | -4.2 (0.73)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Panretinal Photocoagulation Laser Arm; 1; Test type: Non-Inferiority — Non-inferiority of brolucizumab to PRP with respect to change from baseline in BCVA at Week 54, considering a non-inferiority margin of 4 ETDRS letters. Assuming that the BCVA changes follow a normal distribution with equal means between treatments, and a common standard deviation of 10 letters, for a one-sided alpha level of 0.025, with 300 subjects per arm there is >99% power to reject the null hypothesis that brolucizumab 6 mg is inferior to PRP; p < 0.001, ANCOVA; LS mean difference = 4.4, 95% CI 2-sided [2.4 to 6.4], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Panretinal Photocoagulation Laser Arm; 2; Test type: Superiority; p < 0.001, ANCOVA

2. Secondary Outcome: Number and Percentage of Subjects With no Proliferative Diabetic Retinopathy (PDR) at Week 54 for the Study Eye
Description: Proliferative diabetic retinopathy (PDR) is derived from the diabetic retinopathy severity scale (DRSS) as assessed by the central reading center (CRC) using 7-field color fundus photography image. The DRSS on the original score with scores varying from 10 (DR absent) to 85 (very advanced PDR) were then converted into a 12-level scale (Range is from 1 - diabetic retinopathy (DR) absent, to 12- very advanced PDR). (A lower score represents a better outcome.) The event of "No PDR" is then defined as DRSS (12-level scale) < 7.
Time Frame: Week 54
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 294 | 290
Participants | 187 | 65
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Panretinal Photocoagulation Laser Arm; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in % of Participants = 39.4, 95% CI 2-sided [32.0 to 46.8]

3. Secondary Outcome: Number and Percentage of Subjects With no Proliferative Diabetic Retinopathy (PDR) at Week 96 for the Study Eye
Description: as for outcome 2
Time Frame: Week 96
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 310 | 303
Participants | 188 | 86

4. Secondary Outcome: Number and Percentage of Subjects With Center-involved Diabetic Macular Edema (CI- DME) up to Week 54 for the Study Eye
Description: Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
  PRP = Panretinal photocoagulation laser
Time Frame: Up to Week 54
Population: Full Analysis Set (FAS), for patients with a valid measurement with no protocol deviations with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 347 | 341
Participants | 108 | 248
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Panretinal Photocoagulation Laser Arm; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in % of Participants = -41.1, 95% CI 2-sided [-48.0 to -34.2]

5. Secondary Outcome: Number and Percentage of Subjects With Center-involved Diabetic Macular Edema (CI- DME) up to Week 96 for the Study Eye
Description: as for outcome 4
Time Frame: Up to Week 96
Population: Full Analysis Set (FAS), for patients with a valid measurement with no protocol deviations with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 347 | 341
Participants | 126 | 262

6. Secondary Outcome: Area Under the Curve in Change From Baseline in BCVA up to Week 54 and up to Week 96 - for the Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of >= 34 ETDRS letters (Snellen equivalent 20/200) at Screening / Baseline in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better functioning.
  Last observation carried forward (LOCF) was used for the imputation of missing values.
  The AUC in change from Baseline in BCVA up to Week 54 (or Week 96) is referred to as the averaged change from Baseline in BCVA at each visit up to 54 (or Week 96), which was calculated as (BCVA at Week 6 + BCVA at Week 12 + ... + BCVA at Week 54 (or Week 96)) / number of visits with valid BCVA data from Week 6 to Week 54 (or Week 96) - BCVA at Baseline.
Time Frame: Baseline, up to Week 54 and up to Week 96
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Letters read
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 342 | 337
Letters read
  up to Week 54 | 0.5 [-0.4 to 1.4] | -3.2 [-4.2 to -2.3]
  up to Week 96 | -0.1 [-1.2 to 1.1] | -4.3 [-5.4 to -3.1]

7. Secondary Outcome: Diabetic Retinopathy Severity Scale (DRSS): Number and Percentage of Subjects With ≥2 Steps Improvement From Baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) DRSS Score at Week 54 and Week 96
Description: Severity of Diabetic retinopathy was evaluated using the ETDRS DRSS score assessed by the Central Reading Center based on color fundus photography images in the study eye. When the ETDRS-DR severities were evaluable, they were categorized on the original scale with scores varying from 10 (DR absent) to 85 (very advanced PDR). All DRSS values were then converted into a 12-level scale, allowing the derivation of the ≥2-step and ≥3-step change from baseline for each post-baseline assessment".
  A lower score represents better functioning.
Time Frame: Baseline, Week 54 and Week 96
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 295 | 289
Participants
  Week 54 (n=282, 279): number analyzed (Participants) | 282 | 279
  Week 54 (n=282, 279) | 128 | 57
  Week 96 (n=295, 289) | 123 | 65
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Panretinal Photocoagulation Laser Arm; Week 54; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in % of Participants = 26.4, 95% CI 2-sided [19.5 to 33.3]

8. Secondary Outcome: Diabetic Retinopathy Severity Scale (DRSS): Number and Percentage of Subjects With ≥2 Steps Worsening From Baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) DRSS Score at Week 54 and Week 96
Description: as for outcome 7
Time Frame: Baseline, Week 54 and Week 96
Population: Full Analysis Set- Observed, for patients with a valid measurement with no protocol deviations with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 236 | 220
Participants
  Week 54 (n=225,220): number analyzed (Participants) | 225 | 220
  Week 54 (n=225,220) | 6 | 31
  Week 96 (n=236, 201): number analyzed (Participants) | 236 | 201
  Week 96 (n=236, 201) | 18 | 27

9. Secondary Outcome: Diabetic Retinopathy Severity Scale (DRSS): Number and Percentage of Subjects With ≥3 Steps Improvement From Baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) DRSS Score at Week 54 and Week 96
Description: as for outcome 7
Time Frame: Baseline, Week 54 and Week 96
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 295 | 289
Participants
  Week 54 (n=282, 279): number analyzed (Participants) | 282 | 279
  Week 54 (n=282, 279) | 58 | 30
  Week 96 (n=295, 289) | 49 | 33

10. Secondary Outcome: Diabetic Retinopathy Severity Scale (DRSS): Number and Percentage of Subjects With ≥3 Steps Worsening From Baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) DRSS Score at Week 54 and Week 96
Description: as for outcome 7
Time Frame: Baseline, Week 54 and Week 96
Population: Full Analysis Set-Observed, for patients with a valid measurement with no protocol deviations with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 236 | 220
Participants
  Week 54 (n=225, 220): number analyzed (Participants) | 225 | 220
  Week 54 (n=225, 220) | 4 | 16
  Week 96 (n=236, 201): number analyzed (Participants) | 236 | 201
  Week 96 (n=236, 201) | 11 | 16

11. Secondary Outcome: Number and Percentage of Subjects Developing Vision-threatening Complications Associated With Diabetic Retinopathy up to Week 54 and up to Week 96
Description: The vision-threatening complications associated with Diabetic retinopathy (DR) are defined as any event of the following list occurring in the study eye at any time point after Baseline:
  * Center-involved Diabetic macular edema (CI-DME) as defined as Central sub-field thickness (CSFT) ≥280 µm according to Central reading center (CRC) evaluation of Optical coherent tomography (OCT) image
  * Retinal detachment
  * Vitreous hemorrhage
  * Neovascular glaucoma, iris/ anterior chamber angle neovascularization
  * Vitrectomy for DR complications
Time Frame: up to Week 54 and up to Week 96
Population: Full Analysis Set - Observed, for patients with a valid measurement with no protocol deviations with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 347 | 342
Participants
  up to Week 54 | 117 | 258
  up to Week 96 | 144 | 270

12. Secondary Outcome: Ocular AEs (>= 2% in Any Treatment Arm) by Preferred Term for the Study Eye
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  AEs that started after alternative diabetic retinopathy treatment/relevant diabetic macular edema treatment in the study eye are censored.
Time Frame: Adverse events are reported from first dose of study treatment up to Week 90, plus approximately 6 weeks post-treatment, up to a maximum timeframe of approximately 96 weeks.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 347 | 342
Participants
  Number of subjects with at least one AE | 152 | 199
  -Vitreous hemorrhage | 38 | 83
  -Cataract | 26 | 27
  -Dry eye | 15 | 8
  -Intraocular pressure increased | 12 | 3
  -Conjunctival hemorrhage | 10 | 5
  -Macular oedema | 9 | 34
  -Vitreous floaters | 9 | 9
  -Conjunctivitis | 7 | 4
  -Diabetic retinal oedema | 7 | 36
  -Retinal hemorrhage | 5 | 12
  -Diabetic retinopathy | 4 | 13
  -Eye pain | 3 | 7

13. Secondary Outcome: Non-ocular AEs (≥ 2% in Any Treatment Arm) by Preferred Term
Description: as for outcome 12
Time Frame: as for outcome 12
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Panretinal Photocoagulation Laser Arm
Number analyzed (Participants) | 347 | 342
Participants
  Number of subjects with at least one AE | 226 | 217
  COVID-19 | 44 | 47
  Hypertension | 35 | 24
  Upper respiratory tract infection | 28 | 16
  Nasopharyngitis | 22 | 16
  Anaemia | 15 | 15
  Cough | 15 | 10
  Pyrexia | 15 | 7
  Hyperglycaemia | 13 | 10
  Hyperkalaemia | 12 | 2
  Urinary tract infection | 12 | 13
  Diabetes mellitus | 10 | 5
  Pneumonia | 10 | 4
  Coronary artery disease | 9 | 5
  Hyperlipidaemia | 9 | 8
  Hyperuricaemia | 9 | 4
  Chronic kidney disease | 8 | 5
  Depression | 8 | 3
  Blood glucose increased | 7 | 5
  Hypercholesterolaemia | 7 | 5
  Nausea | 7 | 6
  Type 2 diabetes mellitus | 7 | 6
  Arthralgia | 5 | 7
  Influenza | 5 | 8
  -Vomiting | 5 | 9
  Diabetic neuropathy | 2 | 10
  Diabetic foot | 1 | 7

14. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths are reported from first dose of study treatment until end of study treatment at the time of the interim analysis, plus 4 weeks post treatment, up to a maximum timeframe of approximately 96 weeks. Post-treatment deaths are reported for the timeframe of greater than 30 days after last treatment, also up to Week 96. All deaths refer to the sum of on-treatment and post-treatment deaths.
Time Frame: On-treatment - within 30 days after last treatment, up to Week 96; Post-treatment - greater than 30 days after last treatment, also up to Week 96.
Reporting Status: Not Posted, anticipated posting 9999-08

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment up to Week 90, plus approximately 6 weeks post-treatment, up to a maximum timeframe of approximately 96 weeks.
Description: AEs that started after alternative diabetic retinopathy treatment/relevant diabetic macular edema treatment in the study eye are not censored.
Groups:
- Brolucizumab 6mg: Brolucizumab 6 mg: 3 x q6w loading then q12w maintenance through Week 90, with the option from Week 48 onwards to extend the treatment interval by 6 weeks at a time up to 24 weeks and revert to q12w if disease worsens. More frequent injection with q6w interval in the maintenance phase could be administered at the discretion of the Investigator if the disease worsens.
- Overall: Overall
Arm/Group | Brolucizumab 6mg | Panretinal Photocoagulation Laser Arm | Overall
All-Cause Mortality (participants affected / at risk) | 8/347 | 9/342 | 17/689
Serious Adverse Events (participants affected / at risk) | 96/347 | 105/342 | 201/689
Other Adverse Events (participants affected / at risk) | 241/347 | 254/342 | 495/689
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=347) | Panretinal Photocoagulation Laser Arm (N=342) | Overall (N=689)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Acute cardiac event (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 4 | 4
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 2 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0 | 2
Cardiac failure (Cardiac disorders) | 2 | 0 | 2
Cardiac failure acute (Cardiac disorders) | 2 | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 3 | 2 | 5
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 4 | 5
Myocarditis (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Endocrine pancreatic disorder (Endocrine disorders) | 1 | 0 | 1
Cataract - Fellow eye (Eye disorders) | 2 | 1 | 3
Cataract - Study eye (Eye disorders) | 1 | 4 | 5
Cataract cortical - Study eye (Eye disorders) | 0 | 1 | 1
Diabetic retinopathy - Fellow eye (Eye disorders) | 2 | 1 | 3
Diabetic retinopathy - Study eye (Eye disorders) | 0 | 2 | 2
Epiretinal membrane - Fellow eye (Eye disorders) | 0 | 1 | 1
Glaucoma - Fellow eye (Eye disorders) | 0 | 1 | 1
Glaucoma - Study eye (Eye disorders) | 0 | 3 | 3
Macular hole - Fellow eye (Eye disorders) | 1 | 0 | 1
Macular oedema - Fellow eye (Eye disorders) | 0 | 1 | 1
Macular oedema - Study eye (Eye disorders) | 0 | 2 | 2
Pupillary block - Study eye (Eye disorders) | 0 | 1 | 1
Retinal artery occlusion - Study eye (Eye disorders) | 1 | 0 | 1
Retinal detachment - Fellow eye (Eye disorders) | 1 | 0 | 1
Retinal detachment - Study eye (Eye disorders) | 1 | 0 | 1
Retinal haemorrhage - Fellow eye (Eye disorders) | 1 | 0 | 1
Retinal haemorrhage - Study eye (Eye disorders) | 0 | 1 | 1
Retinal neovascularisation - Fellow eye (Eye disorders) | 1 | 0 | 1
Retinal occlusive vasculitis - Study eye (Eye disorders) | 2 | 0 | 2
Retinal vasculitis - Study eye (Eye disorders) | 1 | 0 | 1
Retinopathy proliferative - Fellow eye (Eye disorders) | 1 | 0 | 1
Strabismus - Fellow eye (Eye disorders) | 1 | 0 | 1
Tractional retinal detachment - Fellow eye (Eye disorders) | 1 | 1 | 2
Tractional retinal detachment - Study eye (Eye disorders) | 2 | 3 | 5
Uveitis - Study eye (Eye disorders) | 3 | 0 | 3
Vitreous haemorrhage - Fellow eye (Eye disorders) | 14 | 9 | 23
Vitreous haemorrhage - Study eye (Eye disorders) | 4 | 19 | 23
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Chest pain (General disorders) | 1 | 1 | 2
Death (General disorders) | 0 | 1 | 1
Generalised oedema (General disorders) | 1 | 1 | 2
Hernia pain (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 2
Abscess limb (Infections and infestations) | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0 | 2
Cellulitis (Infections and infestations) | 2 | 2 | 4
Cellulitis staphylococcal (Infections and infestations) | 0 | 1 | 1
Endophthalmitis - Study eye (Infections and infestations) | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 1
Escherichia infection (Infections and infestations) | 1 | 0 | 1
Gangrene (Infections and infestations) | 1 | 1 | 2
Localised infection (Infections and infestations) | 1 | 1 | 2
Mastitis (Infections and infestations) | 1 | 0 | 1
Measles (Infections and infestations) | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 1 | 3
Otitis media chronic (Infections and infestations) | 0 | 2 | 2
Pitted keratolysis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 2 | 2
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Wound infection (Infections and infestations) | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Hyphaema - Study eye (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood glucose increased (Investigations) | 1 | 1 | 2
Blood potassium increased (Investigations) | 1 | 0 | 1
Blood pressure abnormal (Investigations) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 1
Intraocular pressure increased - Study eye (Investigations) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 5 | 1 | 6
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 4
Coma (Nervous system disorders) | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 2 | 2
Dystonia (Nervous system disorders) | 0 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 2 | 5
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 4 | 5
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 1
End stage renal disease (Renal and urinary disorders) | 1 | 3 | 4
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 3
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 1 | 4
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 4 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 5 | 1 | 6
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 2 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=347) | Panretinal Photocoagulation Laser Arm (N=342) | Overall (N=689)
Anaemia (Blood and lymphatic system disorders) | 15 | 16 | 31
Cataract - Fellow eye (Eye disorders) | 22 | 28 | 50
Cataract - Study eye (Eye disorders) | 26 | 29 | 55
Conjunctival haemorrhage - Study eye (Eye disorders) | 10 | 7 | 17
Diabetic retinal oedema - Fellow eye (Eye disorders) | 20 | 18 | 38
Diabetic retinal oedema - Study eye (Eye disorders) | 8 | 41 | 49
Diabetic retinopathy - Fellow eye (Eye disorders) | 14 | 15 | 29
Diabetic retinopathy - Study eye (Eye disorders) | 4 | 15 | 19
Dry eye - Fellow eye (Eye disorders) | 14 | 9 | 23
Dry eye - Study eye (Eye disorders) | 15 | 11 | 26
Epiretinal membrane - Study eye (Eye disorders) | 7 | 3 | 10
Eye pain - Study eye (Eye disorders) | 3 | 7 | 10
Macular oedema - Fellow eye (Eye disorders) | 9 | 12 | 21
Macular oedema - Study eye (Eye disorders) | 9 | 34 | 43
Retinal haemorrhage - Study eye (Eye disorders) | 5 | 11 | 16
Tractional retinal detachment - Study eye (Eye disorders) | 4 | 7 | 11
Visual acuity reduced - Fellow eye (Eye disorders) | 7 | 4 | 11
Vitreous detachment - Study eye (Eye disorders) | 6 | 7 | 13
Vitreous floaters - Study eye (Eye disorders) | 9 | 9 | 18
Vitreous haemorrhage - Fellow eye (Eye disorders) | 35 | 48 | 83
Vitreous haemorrhage - Study eye (Eye disorders) | 40 | 78 | 118
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 6 | 13
Vomiting (Gastrointestinal disorders) | 4 | 9 | 13
Pyrexia (General disorders) | 16 | 7 | 23
Bronchitis (Infections and infestations) | 4 | 7 | 11
COVID-19 (Infections and infestations) | 44 | 53 | 97
Conjunctivitis - Fellow eye (Infections and infestations) | 8 | 5 | 13
Conjunctivitis - Study eye (Infections and infestations) | 7 | 4 | 11
Influenza (Infections and infestations) | 5 | 8 | 13
Nasopharyngitis (Infections and infestations) | 22 | 17 | 39
Upper respiratory tract infection (Infections and infestations) | 30 | 18 | 48
Urinary tract infection (Infections and infestations) | 11 | 13 | 24
Intraocular pressure increased - Fellow eye (Investigations) | 10 | 3 | 13
Intraocular pressure increased - Study eye (Investigations) | 11 | 5 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 5 | 14
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 7 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 10 | 21
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 3 | 14
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 10 | 20
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 5 | 16
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 7 | 7 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 12
Diabetic neuropathy (Nervous system disorders) | 3 | 9 | 12
Depression (Psychiatric disorders) | 8 | 3 | 11
Chronic kidney disease (Renal and urinary disorders) | 7 | 4 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12 | 27
Hypertension (Vascular disorders) | 31 | 29 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04278417/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT04278417/SAP_001.pdf